CLINICAL TRIAL: NCT02274649
Title: A Patient Centered Approach to Successful Community Transition After Catastrophic Injury: Clinical Trial to Evaluate One-to-one Peer Mentoring
Brief Title: Clinical Trial to Evaluate One-to-one Peer Mentoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Responsible Party: Principal Investigator, Julie Gassaway, Direct Wellness Research, Shepherd Center, Atlanta GA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 581327-1
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Results first posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Injuries, Spinal Cord
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Interviewer collecting outcomes data was not aware of group assignment
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention group receiving one-to-one peer mentoring
  Interventions: Behavioral: one-to-one peer mentoring
- Control (Active Comparator): Control group receiving general peer support
  Interventions: Behavioral: general peer support

INTERVENTIONS:
Behavioral: one-to-one peer mentoring — Each patient received one-to-one peer mentoring each week during rehabilitation and for 90 days post discharge
  Arms: Intervention
Behavioral: general peer support — General (traditional) peer support includes introduction and provision of support services upon request
  Arms: Control

SUMMARY:
The research will examine the effects of enhanced peer mentor interactions on facilitating a successful transition to community living following traumatic spinal cord injury (SCI). Participants in the research will be assigned to either (1) the control group that will receive traditional peer mentor types of interactions or (2) to the intervention group that will receive an enhanced peer mentor program called the One-on-One Initiative. Assignment to one of these two groups will occur randomly on admission to Shepherd Center; the only stratifying criteria is injury level - C6 and above vs. C7 and below.

DETAILED DESCRIPTION:
The Peer Support Program was enhanced by the addition of Shepherd staff mentors and volunteer mentors from the community. The Peer Support Supervisor recruited volunteer peer mentors who are at least 10 months post injury, live within a 50 mile radius of Shepherd Center, and have developed a successful reintegration into community living (employed, manage a family, student, etc.). Volunteers completed Shepherd Center volunteer training and were paid a stipend of $20 per patient interaction.

Each recruited volunteer mentor, along with Shepherd Center peer mentor employees, participated in the Christopher and Dana Reeve Foundation peer support mentor training program to help ensure quality interactions with Shepherd Center patients and understand/practice patient confidentiality awareness. This Foundation provides training on a national level by breaking up the country into eight regions - each with a regional coordinator and training program schedule. The faculty and staff of the University of New Mexico developed and maintain the training and certification program, including the mentor management system. The certification program is a "hybrid" program - a series of on-line modules followed by a one-day on-site session. On-line learning is great for conveying information. It saves time and allows everyone to get that information at their own pace. The one-day training session revisits topics covered in the on-line modules: effective peer mentoring, ethics, communication and resources. It includes breakout groups and group discussions. Benefits of partnering with the Foundation, including providing access to certified peer mentors for patients who live outside the Atlanta area are outlined in the attached document (ReevePeer Partnerships.pdf).

A special training session for Shepherd employees/volunteers involved:

1. Part 1: 3-hour on-line course (notification has been sent to potential mentors by CDRF)
2. Part 2: 6-hour face-to-face training meeting at Shepherd Center on March 10, 2014 These training sessions typically are run on a regional basis, so having the program here at Shepherd saved travel expenses and time for the volunteer participants. The PowerPoint used for the March 10 session is attached.

Subjects in the control group received traditional peer support provided by Shepherd Center currently:

1. Within 5-10 days of admission, the patient is introduced to the peer support team.
2. Patients are seen by peer mentors on a referral basis from therapists, nurses, counselors, or physicians or on request from the patient or family.
3. Patients are made aware of monthly peer support meetings, women's groups and caregiver support groups; participation in these groups is optional for patient and/or family.
4. Patients have access to the SCI Peer Support FaceBook page maintained by the Shepherd Peer Mentors

Subjects in the intervention group (and his/her family) received the enhanced One-on-One initiative:

1. Patient was assigned one primary certified peer mentor and 2-3 supplemental mentors to meet individual patient/family needs (if needed). The Peer Support Supervisor matched certified peer mentors with each patient based on characteristics such as age, date of injury, level of injury, cause of injury, marital status, work status before and after injury, interests, leisure activities, and adaptive equipment utilization. Secondary mentors were used to supplement individual patient/family needs. For example, if guidance is needed regarding airline travel, a peer mentor who has mastered airline travel was consulted if the primary peer mentor did not have this experience.
2. Each patient/family evaluated the interaction with his/her peer mentors. PCORI interviewers facilitated completion of this evaluation. Evaluations were reviewed within one week post completion to modify support provided if indicated and ensure that patient/family needs were met.
3. Patients participated in male and female discussion groups, community dinner, and caregiver dinner sponsored by the peer team. Each meeting includes opportunities for discussion in group settings.These meetings are included in the patients' schedules.
4. Peer mentors provide and organize social networking opportunities on FaceBook (Shepherd SCI peers page), CDRF, SCILife, SPINALpedia, facingdisabilities.com,etc.

On the Shepherd SCI Peers Facebook page, the peer mentor supervisor posts questions posed by patients or community members anonymously and feedback volunteered from any of the >2000 Facebook friends.This is especially helpful for sensitive topics that people may not want to be associated with initiating the question.

Evaluation All study patients were interviewed during the 10th-15th day of their stay at Shepherd Center and completed the Self Efficacy scale. Patients were contacted post via telephone at 3, 30, 90 and 180 days post discharge. At each of these times, they were asked healthcare utilization and Self Efficacy questions.

R

ELIGIBILITY:
Inclusion Criteria:

* • All patients admitted to Shepherd Center for rehabilitation following spinal cord injury and discharged to a community setting

Exclusion Criteria:

* • Not discharged from Shepherd Center
* • Discharged from Shepherd Center to non-community setting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jones, PhD, Principal Investigator — VP Clinical Research

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gassaway J, Jones ML, Sweatman WM, Hong M, Anziano P, DeVault K. Effects of Peer Mentoring on Self-Efficacy and Hospital Readmission After Inpatient Rehabilitation of Individuals With Spinal Cord Injury: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Aug;98(8):1526-1534.e2. doi: 10.1016/j.apmr.2017.02.018. Epub 2017 Mar 23. PMID 28342829

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients admitted to SCI inpatient rehabilitation program from April 1 2014 to April 30, 2015 were recruited.
Pre-assignment Details: If planned discharge location was to non-community location, participants were not assigned to group and excluded from study
Groups:
- Intervention: Intervention group receiving one-to-one peer mentoring. Each patient received 1 hour (approximate) of one-to-one peer mentoring each week during rehabilitation and telephone contact each week for 90 days post discharge
- Control: Control group receiving traditional peer support services, which includesintroduction of peer support and provision of support services upon request
Period: Overall Study
Arm/Group | Intervention | Control
Started | 101 | 93
Completed | 77 | 81
Not Completed | 24 | 12

BASELINE CHARACTERISTICS:
Groups:
- Control: Control group receiving traditional peer support services, which includes introduction of peer support and provision of support services upon request
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 101 | 93 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.50 (16.67) | 40.22 (15.78) | 38.80 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 76 | 67 | 143
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 24 | 44
  White | 79 | 66 | 145
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 101 | 93 | 194
Level of injury: paraplegia or tetraplegia [Count of Participants; unit: Participants]
  Paraplegia | 48 | 45 | 93
  Tetraplegia | 53 | 48 | 101

OUTCOME MEASURES:

1. Primary Outcome: Self-efficacy Scale. It Includes an Adapted Self-efficacy Scale From Chronic Disease Literature Focused on Confidence in Managing Self-care Needs Plus Project-specific Items for Assessment of Confidence Regarding Integration Into Community Life.
Description: The General Self-Efficacy scale (6 items) developed at Stanford University for persons with chronic health conditions was adapted for persons with spinal cord injury. Added to this scale were 5 similarly constructed project-specific self-efficacy items focused on community navigation and accessibility (major focus of peer support program).
  Respondents (via telephone interview) provided a response to each of 11 items using a 10-point Likert scale ranging from 1 (not confident) to 10 (very confident). Item response scores were averaged for the total self-efficacy score. Total scores ranged from 11 to 110 (11 items with 10 response options). Higher scores indicate greater self-efficacy to manage injury conditions.
  Growth Curve Analysis was used to determined significant changes over time in self-efficacy. Initial status coefficients depict where participants begin at the first time point (3 days post discharge) and growth rate coefficients show how participants change over time.
Time Frame: 3 days post rehabilitation discharge through 180 days post discharge
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Intervention
Number analyzed (Participants) | 81 | 77
units on a scale | 7.64 (0.300) | 7.65 (0.210)

2. Primary Outcome: Rehospitalization - Number of Days
Description: Rehospitalization days (number) within 30 days post inpatient rehabilitation discharge
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 81 | 77
days | 0.79 (3.19) | 0.49 (2.26)

3. Primary Outcome: Rehospitalization - Percent of Patients Rehospitalized
Description: Percent of patients rehospitalized at 30 days post discharge from inpatient rehabilitation
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | Control | Intervention
Number analyzed (Participants) | 81 | 77
percentage of patients | 9 | 8

4. Secondary Outcome: Rehospitalization - Number of Days (Cumulative)
Description: Rehospitalization days (cumulative) within 90 days post inpatient rehabilitation discharge
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 81 | 77
days | 2.11 (5.42) | 0.99 (4.06)

5. Secondary Outcome: Rehospitalization - Percent of Patients Rehospitalized (90 Days)
Description: Percent of patients (cumulative) rehospitalized within 90 days post discharge from inpatient rehabilitation
Time Frame: 90 days
Measure: Number; unit: percentage of patients
Arm/Group | Control | Intervention
Number analyzed (Participants) | 81 | 77
percentage of patients | 19 | 10

6. Secondary Outcome: Rehospitalization - Number of Days (Cumulative)
Description: Rehospitalization days (cumulative) within 180 days post inpatient rehabilitation discharge
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Intervention
Number analyzed (Participants) | 81 | 77
days | 2.85 (6.54) | 1.55 (5.14)

7. Secondary Outcome: Rehospitalization - Percent of Patients (180 Days)
Description: Percent of patients (cumulative) rehospitalized within 180 days post discharge from inpatient rehabilitation
Time Frame: 180 days
Measure: Number; unit: percentage of paients
Arm/Group | Control | Intervention
Number analyzed (Participants) | 81 | 77
percentage of paients | 22 | 14

ADVERSE EVENTS:
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/81
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/81
Other Adverse Events (participants affected / at risk) | 0/77 | 0/81

LIMITATIONS AND CAVEATS:
Control group received requested peer support services; may have contributed to the relatively modest effect size. We cannot claim use of validated measure of self-efficacy; we adapted a measurement validated in other populations and added items.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No